CLINICAL TRIAL: NCT04047576
Title: Prospective Study of Prednisone Versus Sirolimus in the Treatment of Idiopathic Retroperitoneal Fibrosis
Brief Title: Study of Sirolimus in Idiopathic Retroperitoneal Fibrosis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peking University International Hospital (Other)
Responsible Party: Principal Investigator, Gao Hui, Principal Investigator, Peking University International Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sirolimus for RPF
Record Dates: First submitted 2019-07-25; First posted 2019-08-06 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Retroperitoneal Fibrosis
Keywords: mTOR inhibitor; Sirolimus; Retroperitoneal Fibrosis
MeSH Terms: conditions — Retroperitoneal Fibrosis | interventions — Sirolimus; Adrenal Cortex Hormones; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sirolimus group (Experimental): Sirolimus: 2 mg/day for the first 3 days and 1 mg/day thereafter. The plasma drug concentration was monitored at 14 days, 12 weeks, and 48 weeks of medication to maintain a plasma drug concentration of 4-15 ug/L.
  Prednisone: 0.8 mg/kg/d (maximum dose: 60 mg/d), reduced by 5 mg every 14 days, by 2.5 mg every 2 weeks after 30 mg/d until discontinuation.
  Interventions: Drug: Sirolimus; Drug: Corticosteroid
- corticosteroid group (Active Comparator): Prednisone: 0.8 mg/kg/d (maximum dose: 60 mg/d), reduced by 5 mg every 14 days, by 2.5 mg every 2 weeks after 30 mg/d until 5-7.5 mg/d.
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Drug: Sirolimus — The efficacy is evaluated at 12 weeks, and treatment will be adjusted according to the control of disease and adverse effects.For experimental group, if a patient is assessed as treatment failure (TS), the patient should be withdrawn from the study and receive rescue treatment. Whereas, a patient would be transferred to the control group if he/ she cann't stand the side effects of sirolimus but not serious adverse event (SAE).
  Arms: sirolimus group
Drug: Corticosteroid — The efficacy is evaluated at 12 weeks, and treatment will be adjusted according to the control of disease and adverse effects. For active comparator group, if a patient is assessed as treatment failure (TF), the patient should be withdrawn from the study and receive rescue treatment.
  Other Names: Prednisone

SUMMARY:
Retroperitoneal fibrosis refers to a group of diseases characterized by hyperplasia of the fibrosclerotic tissues in the retroperitoneal space, which can compress the surrounding ureters and inferior vena cava and cause serious complications such as aortic aneurysm, renal failure, and even death. The lesion is diffuse and difficult to resect. corticosteroid is the first-line medication, but the recurrence rate of the disease is high, especially after dose reduction of corticosteroid. Therefore, the combined use of immunosuppressants is very important in preventing disease recurrence and reducing the toxic and side effects of long-term corticosteroid. Sirolimus plays dual roles in inhibiting lymphocyte activation and fibroblast proliferation. It is inferred from its mechanism that sirolimus is a good potential treatment option for idiopathic retroperitoneal fibrosis. Therefore, we conducted this RCT on patients with idiopathic retroperitoneal fibrosis to determine the efficacy and safety of sirolimus.

DETAILED DESCRIPTION:
Retroperitoneal fibrosis refers to a group of diseases characterized by hyperplasia of the fibrosclerotic tissues in the retroperitoneal space, which mostly involve the abdominal aorta and iliac artery distal to the kidneys. The hyperplastic tissues can compress the surrounding ureters and inferior vena cava and cause serious complications such as aortic aneurysm, renal failure, and even death. There is no clear boundary between the lesion and its surrounding tissues. The lesion is diffuse and difficult to resect. corticosteroid is the first-line medication, but the recurrence rate of the disease is high, especially after dose reduction of corticosteroid. Therefore, the combined use of immunosuppressants is very important in preventing disease recurrence and reducing the toxic and side effects of long-term high- and medium-dose corticosteroid. In recent years, as the immunological characteristics of retroperitoneal fibrosis have gradually been recognized, some rheumatologists and immunologists have attempted to use immunosuppressants commonly used for autoimmune diseases in this population, including biologics. However, high-level evidences of evidence-based medicine such as randomized controlled trials (RCTs) were still lacking. Sirolimus plays dual roles in inhibiting T lymphocyte activation and fibroblast proliferation. It is inferred from its mechanism that sirolimus is a good potential treatment option for idiopathic retroperitoneal fibrosis. Therefore, we conducted this RCT on patients with idiopathic retroperitoneal fibrosis to determine the efficacy and safety of sirolimus.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic retroperitoneal fibrosis diagnosed on CT or MRI. For patients with suspected secondary retroperitoneal fibrosis or atypical idiopathic retroperitoneal fibrosis suggested by imaging, idiopathic retroperitoneal fibrosis should be confirmed by puncture biopsy
2. Increased ESR and CRP levels caused by this disease and/or active lesions suggested on imaging

Exclusion Criteria:

1. Secondary retroperitoneal fibrosis
2. Having used corticosteroid (equivalent to >10 mg per day of prednisone), immunosuppressant, or biologic within 3 months prior to enrollment
3. Having any contraindication of prednisone or sirolimus, or allergy to sirolimus, or having experienced serious adverse reactions from the previous use of any of the above drugs
4. Massive proteinuria (24-hour urine protein quantitation ≥3 g), moderate-to-severe anemia (hemoglobin <90 g/L), agranulocytosis (white blood cell count <1.5×10^9/L or neutrophil count <0.5×10^9/L), platelet count <50×10^9/L, interstitial pneumonia
5. Uncontrollable diabetes, hypertension, hyperlipidemia, infection, or heart failure, or other serious complications
6. Malignancy
7. Pregnancy or need for pregnancy in the near future
8. Unable to adhere to follow-up or refuses to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Treatment failure rate | 12 weeks of treatment
Cumulative dose of prednisone | 48 weeks
Size of retroperitoneal fibrotic mass | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hui Gao, Doctor, Principal Investigator — Peking University International Hospital
Locations (1):
- Peking University International Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No